CLINICAL TRIAL: NCT01227005
Title: Early Whole Blood in Patients Requiring Transfusion After Major Trauma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bryan Cotton, Associate Professor, Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-07-1-0229
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Trauma/Injury Problem
Keywords: Transfusion; Whole Blood; Trauma; Coagulopathy; Component Therapy; Civilian; Military
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries; Hemostatic Disorders | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole Blood (Active Comparator): Whole Blood plus pooled platelets
  Interventions: Biological: Transfusion of blood products
- Component Therapy (Active Comparator): Red blood cells, plasma, platelets
  Interventions: Biological: Transfusion of blood products

INTERVENTIONS:
Biological: Transfusion of blood products — The intervention will be either a) administration of 1 unit of whole blood plus pooled products or b) administration of component therapy (red blood cells, plasma, platelets).

SUMMARY:
The proposal will assess if patients who require massive transfusion can be accurately predicted early after emergency department arrival and assess if the use of stored whole blood during initial resuscitation will reduce transfusion needs compared to transfusion with component therapy and thus improve outcome.

DETAILED DESCRIPTION:
Background: The acquired coagulopathy of trauma is responsible for a large percentage of early deaths in civilian trauma practice and is a major cause of battlefield mortality. Widespread recognition has provided a rationale for fundamental changes in the initial management of severely injured patients through prevention of hypothermia, damage control surgery, massive transfusion protocols and early triage to intensive care units for optimized resuscitation. Despite these major advances, hemorrhage remains a leading cause of early death in both civilian trauma and military combat casualty care. However, it is unclear how early whole blood will affect coagulopathy in this cohort of patients as compared to the current standard of care. Objective/Hypothesis: The proposal will assess if patients who require massive transfusion can be accurately predicted early after emergency department arrival and assess if the use of stored whole blood during initial resuscitation will reduce transfusion needs compared to transfusion with component therapy and thus improve outcome.

Study Design: As a first step in testing this hypothesis, we will test commonly utilized point of care analysis devices and determine their reliability in predicting transfusion requirements in severely injured trauma patients within 20 minutes after arrival in the emergency department. Furthermore, we will prospectively randomize severely injured patients who require a blood transfusion to receive either stored whole blood and pooled platelets or component therapy (packed red blood cells, fresh frozen plasma, and platelets, our current standard of care) and compare the ability of stored whole blood to reduce transfusion needs and improve clinical outcomes.

Relevance: Severe uncontrollable coagulopathy in major trauma patients continues to be a major determinant of trauma mortalities. The proposed effort aims to provide an early, coagulopathy-based prediction model to identify patients at risk for massive transfusion. Moreover, our proposal intends to evaluate early stored whole blood transfusion in this at risk patient population and determine stored whole blood's ability to prevent or control severe coagulopathy compared to standard transfusion care.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Meet Code 3 status; Code 3 is determined by the following criteria (Patients must meet at least one of the following physiologic and/or anatomic criteria):

   * Physiologic criteria indicating high risk or life threatening injuries
   * GCS <10 (Glasgow Coma Scale)
   * SBP <90 (Systolic blood pressure)
   * RR <10 or >29 (Respiratory rate)
   * HR >120 (Heart rate)
   * intubated
   * Base Deficit > 6
   * Anatomic criteria indicating high risk or life threatening injuries
   * Any penetrating injury to torso, groin, or neck
   * Amputation proximal to the ankle or wrist
   * Uncontrolled external hemorrhage
   * Two or more long bone fractures
   * Pelvic fracture
   * Paraplegia or quadriplegia
   * Combination trauma with burns ≥ 20% BSA (body surface area)
3. Demonstrate evidence of blood loss due to injury, requiring transfusion in the ED.

Exclusion Criteria:

1. Death thought to be imminent, suggesting a futile resuscitation effort
2. Known or assumed religious objection to blood products
3. Do not resuscitate order in place
4. Women who present to the ED who are obviously pregnant.
5. Patients who appear to the ED wearing the -opt-out‖ bracelet provided at the community consultation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Cotton, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital - Texas Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] Erber WN, Tan J, Grey D, Lown JA. Use of unrefrigerated fresh whole blood in massive transfusion. Med J Aust. 1996 Jul 1;165(1):11-3. doi: 10.5694/j.1326-5377.1996.tb124809.x. PMID 8676771
- [Background] Mohr R, Martinowitz U, Lavee J, Amroch D, Ramot B, Goor DA. The hemostatic effect of transfusing fresh whole blood versus platelet concentrates after cardiac operations. J Thorac Cardiovasc Surg. 1988 Oct;96(4):530-4. PMID 3172799
- [Background] Oberman HA. The indications for transfusion of freshly drawn blood. JAMA. 1967 Jan 9;199(2):93-7. No abstract available. PMID 5333702
- [Background] Grosso SM, Keenan JO. Whole blood transfusion for exsanguinating coagulopathy in a US field surgical hospital in postwar Kosovo. J Trauma. 2000 Jul;49(1):145-8. doi: 10.1097/00005373-200007000-00022. PMID 10912871
- [Background] Ledgerwood AM, Lucas CE. A review of studies on the effects of hemorrhagic shock and resuscitation on the coagulation profile. J Trauma. 2003 May;54(5 Suppl):S68-74. doi: 10.1097/01.TA.0000064513.59253.70. PMID 12768106
- [Derived] Cotton BA, Podbielski J, Camp E, Welch T, del Junco D, Bai Y, Hobbs R, Scroggins J, Hartwell B, Kozar RA, Wade CE, Holcomb JB; Early Whole Blood Investigators. A randomized controlled pilot trial of modified whole blood versus component therapy in severely injured patients requiring large volume transfusions. Ann Surg. 2013 Oct;258(4):527-32; discussion 532-3. doi: 10.1097/SLA.0b013e3182a4ffa0. PMID 23979267

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Whole Blood | Component Therapy
Started | 55 | 52
Completed | 50 | 51
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Whole Blood | Component Therapy | Total
Number analyzed (Participants) | 55 | 52 | 107
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [29 to 56] | 38 [32 to 56] | 39 [30 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 43 | 43 | 86
Region of Enrollment [Number; unit: participants]
  United States | 55 | 52 | 107

OUTCOME MEASURES:

1. Primary Outcome: Units of Blood Products Required During the First 24 Hours After Emergency Department Admission
Description: Compare the ability of whole blood to reduce initial 24-hour transfusion requirements as compared to component therapy (red blood cells, plasma, and platelet units)
Time Frame: first 24 hours after ED admission
Measure: Median (Inter-Quartile Range); unit: units of blood
Arm/Group | Whole Blood | Component Therapy
Number analyzed (Participants) | 55 | 52
units of blood | 12 [6 to 24] | 13 [5 to 29]

2. Secondary Outcome: 24-hour Mortality
Description: Mortality rate at 24 hours after arrival
Time Frame: First 24 hours after ED admission
Measure: Number; unit: participants
Arm/Group | Whole Blood | Component Therapy
Number analyzed (Participants) | 55 | 52
participants | 12 | 7

3. Secondary Outcome: 30-day Mortality
Description: Evaluate 30-day mortality among those receiving whole blood compared to those receiving component therapy
Time Frame: first 30 days after ED admission
Measure: Number; unit: participants
Arm/Group | Whole Blood | Component Therapy
Number analyzed (Participants) | 55 | 52
participants | 15 | 8

ADVERSE EVENTS:
Arm/Group | Whole Blood | Component Therapy
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/52
Other Adverse Events (participants affected / at risk) | 1/55 | 0/52
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole Blood (N=55) | Component Therapy (N=52)
Allergic reaction to blood product (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Allergic reaction to blood product in WB arm.

LIMITATIONS AND CAVEATS:
First, we failed to specifically exclude patients with severe TBI from our initial protocol. Finally, we did not use an objective scoring system to randomize patients and, therefore, did not always include patients who would have received an MT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No